CLINICAL TRIAL: NCT05452252
Title: Functional Mandibular Evaluation and Anthropometric Facial Analysis In Relation With Neck Profile In Adolescents With İdiopathic Scoliosis
Brief Title: Mandibular Evaluation and Facial Analysis In Adolescents With Idiopathic Scoliosis
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Fatih Çelik, PhD(s), Hacettepe University
Other Study IDs: GO20/694
Record Dates: First submitted 2022-07-06; First posted 2022-07-11 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Scoliosis Idiopathic
Keywords: Scoliosis; Temporomandibular Joint; Facial Asymmetry; Neck
MeSH Terms: conditions — Scoliosis; Facial Asymmetry

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- study group: adolescents with idiopathic scoliosis
  Interventions: Diagnostic Test: functional mandibular evaluation
- control group: healthy individuals
  Interventions: Diagnostic Test: functional mandibular evaluation

INTERVENTIONS:
Diagnostic Test: functional mandibular evaluation — Active mandibular movements including depression, protrusion, and left-right deviation, facial anthropometry was measured on facial shape on photograph, and phenotype and asymmetry
  Other Names: anthropometric facial analysis

SUMMARY:
Fifty-eight participants with AIS and 45 healthy controls were included in the study. Active mandibular movements including depression, protrusion, and left-right deviation were assessed with a ruler. Facial anthropometry was measured on facial shape on photograph, and phenotype and asymmetry were determined from the acquired anthropometric facial data. Neck mobility was evaluated in movements of flexion, extension, right-left lateral flexion, and right-left rotation using a standard flexible tape. The Fremantle Neck Awareness Questionnaire was used to assess neck awareness. Neck pain in the previous week was measured with a Visual Analog Scale.

DETAILED DESCRIPTION:
Functional evaluation of the mandible was performed by measuring active mandibular movements (Fig 1). For mandibular depression, participants were asked to open their mouths as much as they could without pain. The distance between central incisors of the mandibular row of teeth and the maxillary row of the obturator was recorded. For mandible protrusion, they pushed their lower jaws forward as far as they could and the distance between the upper and lower jaws were recorded. For mandibular deviation, participants pushed their lower jaws first left and then right, and lateral mandibular excursions were measured from upper incisal midline to lower midline. All measurements were performed with the help of a 20-cm ruler and recorded in cm 16.

Facial anthropometry was measured on photograph. A digital camera mounted on a tripod at 110 centimeters in height and a distance of 100 centimeters was used to take photographs 17. Participants' position was standardized on a previously marked cross on the floor. Those who wear glasses were asked to remove the glasses, and the participants with long hair were asked to tie their hair from the top. They were asked to assume a relaxed standing position when the photographs were taken. A small white square sticker 2 cm × 2 cm was placed on the forehead and on the flat surfaces of the right and left cheeks, with the camera lens perpendicular to the square. The purpose of the sticker was to be able to express linear measurements as centimeters rather than pixels while measuring the 3 sides of facial anthropometric landmarks using the Image J program 18. All participants were photographed at front and right and left sides. The measured anthropometric variables were as follows: physiognomic face height, morphological face height, lower face height, face width, mandible width, right upper facial depth, left upper facial depth, right lower facial depth, left lower facial depth, right midfacial depth, left midfacial depth, biocular width, cheek width (distance between inferior insertion of ear), and mouth width. Landmarks are shown and measured variables are defined in Fig 2 19,20. Face golden ratio was used to determine face shape and facial index was used for face phenotype. Face golden ratio was the ratio of physiognomic facial height to the face width, and facial index was the ratio of morphological face height and maximum face width.

ELIGIBILITY:
Inclusion Criteria:

* 10-18 years old patients
* Cobb's angle of above 10°
* Age-matched healthy group of girls

Exclusion Criteria:

* congenital scoliosis
* spinal deformity
* undergone surgical correction of the spine
* tumor
* rheumatological disease
* neuromuscular disease
* cardiovascular disease
* pulmonary disease
* renal disease
* facial surgery
* dental treatments

Ages: 10 Years to 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — only females included to study
Study Population: 103 adolescents, 58 of them with idiopathic scoliosis and 45 of them healthy, were included in the study.
Sampling Method: Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
mandibular protrusion | 1 day
  mandibular position change due to scoliosis

SECONDARY OUTCOMES:
facial asymmetry | 1 day
  face asymmetry due to scoliosis

CONTACTS AND LOCATIONS:
Overall Officials: fatih çelik, MSc, Study Director — PhD student
Locations (1):
- Fatih Çelik, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided